CLINICAL TRIAL: NCT04042727
Title: Controlling Rapid Atrial Fibrillation With Dexmedetomidine (C-RAD) Trial
Brief Title: Controlling Rapid Atrial Fibrillation With Dexmedetomidine
Acronym: C-RAD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Futility, as a result of COVID-19 impact
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Andreas Kalogeropoulos, Director, Cardiovascular Research, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2019-00250
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Rapid Atrial Fibrillation; Heart Rate Control
Keywords: Dexmedetomidine; Critical Care; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to receive either Dexmedetomidine or Placebo in addition to Standard of Care. Investigational pharmacy will be primarily responsible for randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine plus Standard of Care (Experimental): Dexmedetomidine hydrochloride infusion will be prepared by the investigational pharmacy and administered intravenously at a rate of 1mcg/kg/hr for a duration of 8 hrs to patients in rapid Afib in addition to the usual standard of care as deemed necessary by patient's ICU team.
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Placebo plus Standard of Care (Placebo Comparator): Normal Saline solution will be prepared by investigational pharmacy and administered intravenously at a rate of 1mcg/kg/hr for a duration of 8 hrs to patients in rapid Afib in addition to the usual standard of care as deemed necessary by patient's ICU team.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Six vials of Dexmedetomidine hydrochloride 100mcg/ml (2ml per vial) will be added to a 250mL bag of normal saline by the investigational pharmacy to prepare for infusion by patient's bedside nurse. Infusion rate will be 1mcg/kg/hr.
  Other Names: Precedex
  Arms: Dexmedetomidine plus Standard of Care
Other: Normal Saline — 0.5% sodium chloride (NaCl). The investigational pharmacy will prepare the normal saline placebo 250mL bag for infusion by patient's bedside nurse. Infusion will be 1mcg/kg/hr.
  Other Names: Sodium Chloride Injection
  Arms: Placebo plus Standard of Care

SUMMARY:
The purpose of this study is to assess the effects of Dexmedetomidine (DEX), on heart rate control in patients with rapid atrial fibrillation (AF) through a pragmatic, randomized, double blinded study comparing the addition of Dex or placebo to standard of care (SOC) treatment.

DETAILED DESCRIPTION:
Dexmedetomidine is a commonly used sedative/anxiolytic agent in the ICU with sympatholytic properties that can cause a decrease in heart rate. Eligible patients will be randomized into one of two groups: SOC plus Dex arm or SOC plus placebo (normal saline) arm. Study drug infusion will be administered at an infusion rate of 1μg/kg/hr via IV, and will not include a loading dose. Four 6-second telemetry rhythm strips will be collected per hour, starting one hour prior to study drug infusion, during the eight hour infusion period, and two hours post infusion cessation). Degree of heart rate control and time to heart rate control for both groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients in a SBU Hospital ICU with rapid-AF (with ventricular rates >100 bpm).
* Patient screening will be conducted prior to patient or LAR consent.

Exclusion Criteria:

* Patients age <18yrs;
* Anticipated ICU stay <11hrs;
* Permanently paced heart rhythm;
* Known 2nd or 3rd degree heart block;
* Junctional rhythms;
* Known pregnancy;
* Known allergy to Dexmedetomidine;
* Receiving Dexmedetomidine prior to study onset;
* Non-intubated patients w/ Glasgow Coma Scale <8;
* Weight >400lbs (protocol dosing restriction);
* Untreated, symptomatic hypotension (SBP<90mmHg);
* Received amiodarone, lidocaine, or mexiletine w/in 4hrs prior to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kalogeropoulos, MD MPH PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment has stopped because of challenges associated with the COVID-19 pandemic
Period: Overall Study
Arm/Group | Dexmedetomidine Plus Standard of Care | Placebo Plus Standard of Care
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine Plus Standard of Care | Placebo Plus Standard of Care | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (19.3) | 72.3 (5.15) | 70.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Systolic Blood Pressure
Description: Assess mean systolic blood pressure measurements between the two arms
Time Frame: During Study Drug Infusion Period
Population: Data not collected because of protocol termination
Arm/Group | Dexmedetomidine Plus Standard of Care | Placebo Plus Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24h
Arm/Group | Dexmedetomidine Plus Standard of Care | Placebo Plus Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT04042727/Prot_SAP_000.pdf